CLINICAL TRIAL: NCT02280252
Title: Response, Resistance and Metastasis of Locally Advanced Breast Cancer (LABC, Stage 2B-3C) in a Multiethnic Cohort: A Phase II International Multicentric Study of Concurrent Paclitaxel and Radiation
Brief Title: Study of Concurrent Paclitaxel and Radiation: Correlation of Tumor Profiles With Pathologic Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-209
Record Dates: First submitted 2014-10-08; First posted 2014-10-31 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
Keywords: Locally-advanced Breast Cancer; LABC; breast cancer; breast; cancer; metastasis; metastatic; tumor; radiation; radiation therapy; radiotherapy; paclitaxel
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Paclitaxel; Albumin-Bound Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Concurrent Paclitaxel and RT (Experimental): Patients will be administered pre-operatively over 12 weeks either:
  1. Paclitaxel, 30mg/m^2 twice per week, intravenously over 1 hour on a Monday/Thursday or Tuesday/Friday schedule
  2. Abraxane, 30mg/m^2 twice per week, intravenously administered over 30 minutes, on a Monday/Thursday or Tuesday/Friday schedule
  Patients will concurrently receive 6 weeks of radiation therapy, weeks 2-7:
  Patients will receive a total dose to the breast, axilla and supraclavicular area of 45 Gy at 1.8 Gy/fraction, +14 Gy to the area of the original palpable tumor at 2 Gy/fraction (32 fractions)
  Interventions: Drug: Paclitaxel; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel (including Abraxane), 30 mg/m2 twice per week. Paclitaxel will be given IV over 1 hour, Abraxane® will be administered over 30 min, and administered on a Monday/Thursday or Tuesday/Friday schedule.
  Other Names: Abraxane
Radiation: Radiation therapy — Patients will receive a total dose of 45 Gy to the breast, axilla and supraclavicular area at 1.8 Gy/fraction, +14 Gy to the original palpable tumor at 2 Gy/fraction (total 32 fractions)
  Other Names: radiotherapy

SUMMARY:
The need to understand LABC is especially compelling in populations and countries with limited resources, where breast cancer incidence is relatively low, but mortality is comparably high. In these settings access to appropriate cancer care is characteristically limited or often plainly nonexistent. In contrast to economically developed nations, where on average fewer than 20% of women present with breast cancer at advanced stages, LABC and metastatic disease are the most common stages at presentation in 50% or more women in Latin America, Asia and Africa.

DETAILED DESCRIPTION:
The term -locally advanced breast cancer (LABC) commonly includes tumors whose maximum diameter is 5 cm (T3) or larger, or which present with involvement of the chest wall or skin. Surprisingly, the simultaneous presence of clinically detectable distant metastases is relatively infrequent (~8%), a peculiar finding since in 73% of these large tumors it is possible to document shedding of tumor cells into the blood.

While LABC has become a rare clinical presentation of breast cancer in the general population as a result of improved early detection by mammographic screening, it remains relatively common among minority women of low socioeconomic status. For instance, in a consecutive series of 363 African-American women presenting in a large urban hospital, one out of three women newly diagnosed with breast cancer had LABC.

It is well documented that although the incidence of breast cancer among African-Americans is lower than among white women, breast cancer mortality in African-Americans is significantly higher. In 1998, the American Cancer Society, the National Cancer Institute and the Centers for Disease Control and Prevention reported an overall downward trend in cancer incidence and mortality between 1990 and 1995 for all cancers combined. Many minority and medically underserved populations, however, did not share equally in these improvements. These patients have continued to encounter multifactorial barriers to early detection and care, warranting interventions to improve access.

At the same time, it is equally important to offer the best chance for survival to those underserved women who have already availed themselves of medical care. Paradoxically, while the medical community is aware of the inadequate accrual of minority patients to clinical trials, only few trials exist for LABC.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven locally-advanced breast cancer: IIB, IIIA, and IIIB
* Metastatic breast cancer: limited to the subset of patients with intact breast, locally advanced tumor and involved ipsilateral supraclavicular nodes
* Measureable disease required
* Adequate laboratory values:

Hgb > 10 ANC > 1500 Platelets > 150,000 Creatinine < 1.5 Liver function < 3x normal

* Patient ≥ 18 years of age
* Medically and psychologically able to comply with all study requirements
* ECOG performance score 0-1
* CT chest, abdomen, and pelvis performed
* Mammogram or USG performed
* Signed informed consent

Exclusion Criteria:

* Breast cancer patients with Stage 0, Stage I, or Stage IIA
* Previous XRT or chemotherapy
* Presence of distant metastases documented clinically or radiographically with the exception of ipsilateral supraclavicular nodes
* Pregnancy
* Inflammatory breast cancer
* Patients under treatment (or who will have recently been treated) with anti-neoplastic, immunosuppressive or hormonal medications
* Patients who are found to have a cancer positive for the marker HER-2/neu (applies only to NYU Tisch and Bellevue sites)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2005-03; Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Huppert, M.D., Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The PI and study team has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available
Groups:
- Concurrent Paclitaxel and RT: Patients will be administered pre-operatively over 12 weeks either:
  1. Paclitaxel, 30mg/m^2 twice per week, intravenously over 1 hour on a Monday/Thursday or Tuesday/Friday schedule
  2. Abraxane, 30mg/m^2 twice per week, intravenously administered over 30 minutes, on a Monday/Thursday or Tuesday/Friday schedule
  Patients will concurrently receive 6 weeks of radiation therapy, weeks 2-7:
  Patients will receive a total dose to the breast, axilla and supraclavicular area of 45 Gy at 1.8 Gy/fraction, +14 Gy to the area of the original palpable tumor at 2 Gy/fraction (32 fractions)
  Paclitaxel: Paclitaxel (including Abraxane), 30 mg/m2 twice per week. Paclitaxel will be given IV over 1 hour, Abraxane® will be administered over 30 min, and administered on a Monday/Thursday or Tuesday/Friday schedule.
  Radiation therapy: Patients will receive a total dose of 45 Gy to the breast, axilla and supraclavicular area at 1.8 Gy/fraction, +14 Gy to the original palpable tumor at 2 Gy/fraction (total 32 fractions)
Period: Overall Study
Arm/Group | Concurrent Paclitaxel and RT
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The PI and study team has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available
Arm/Group | Concurrent Paclitaxel and RT
Number analyzed (Participants) | 0
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Study-Specific Measure

OUTCOME MEASURES:

1. Primary Outcome: Test the Clinical Effectiveness of Concurrent Paclitaxel and Radiation in a Multiethnic Cohort
Description: Test the effectiveness of concurrent paclitaxel and radiation in a prospective multiethnic cohort of patients with newly diagnosed stage 2B-3C breast cancer treated at three international academic centers under uniform conditions. Local recurrence, regional recurrence and overall survival will be measured
Time Frame: 4.5 years
Population: as for baseline characteristics
Arm/Group | Concurrent Paclitaxel and RT
Number analyzed (Participants) | 0

2. Secondary Outcome: Measure the Pathological Response Rate of Concurrent Paclitaxel-radiation
Description: Measure the pathological response rate to concurrent paclitaxel-radiation at each collaborating institution and compare it to that achieved in a previous Phase I-II trial
Time Frame: 4.5 years
Population: as for baseline characteristics
Arm/Group | Concurrent Paclitaxel and RT
Number analyzed (Participants) | 0

3. Secondary Outcome: Perform Molecular Biology and Genomic Studies of Obtained Core Biopsies to Identify Biomarkers for Predisposition to Breast Cancer
Description: Obtain core biopsies of the original tumor before and after treatment (from the surgical specimen) for molecular biology and genomic studies of biomarkers and genetic anomalies that may signal a population's predisposition to breast cancer and/or susceptibility to study intervention
Time Frame: 4.5 years
Population: as for baseline characteristics
Arm/Group | Concurrent Paclitaxel and RT
Number analyzed (Participants) | 0

4. Secondary Outcome: Patient Demographics
Description: Acquire descriptive information on patient epidemiological, cultural and behavioral characteristics
Time Frame: 4.5 years
Population: as for baseline characteristics
Arm/Group | Concurrent Paclitaxel and RT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The PI and study team has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Arm/Group | Concurrent Paclitaxel and RT
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT02280252/Prot_SAP_000.pdf